CLINICAL TRIAL: NCT00696228
Title: High Fat Diet: Oxidative Effects and Cardiovascular Risk
Brief Title: High Fat Diet: Oxidative and Cardiovascular Effects
Acronym: AFN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Robert C. Atkins Foundation (Other)
Responsible Party: Principal Investigator, Heidi J. Silver, Research Associate Professor, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 071325
Record Dates: First submitted 2008-06-09; First posted 2008-06-12 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- AFN A (Placebo Comparator): High Fat Diet Placebo
  Interventions: Dietary Supplement: Placebo
- AFN B (Experimental): MUFA
  Interventions: Dietary Supplement: MUFA
- AFN C (Experimental): PUFA
  Interventions: Dietary Supplement: PUFA
- AFN D (Experimental): SFA
  Interventions: Dietary Supplement: SFA

INTERVENTIONS:
Dietary Supplement: Placebo — Placebo
  Arms: AFN A
Dietary Supplement: MUFA — MUFA
  Arms: AFN B
Dietary Supplement: PUFA — PUFA
  Arms: AFN C
Dietary Supplement: SFA — SFA
  Arms: AFN D

SUMMARY:
To test the effects of a modified Atkins high fat diet on endothelial function, insulin resistance and energy balance.

DETAILED DESCRIPTION:
To test the effects of a modified Atkins high fat diet on endothelial function, insulin resistance and energy balance.

ELIGIBILITY:
Inclusion Criteria:

* BMI 30-39.9
* Female
* Age 21-40

Exclusion Criteria:

* Smoker
* Comorbid Disease

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Actual)
Dates: Start 2008-08; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
endothelial function | 4 months

SECONDARY OUTCOMES:
energy balance and body composition | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Heidi J Silver, PhD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Niswender KD, Fazio S, Gower BA, Silver HJ. Balanced high fat diet reduces cardiovascular risk in obese women although changes in adipose tissue, lipoproteins, and insulin resistance differ by race. Metabolism. 2018 May;82:125-134. doi: 10.1016/j.metabol.2018.01.020. Epub 2018 Jan 31. PMID 29382504
- [Derived] Silver HJ, Kang H, Keil CD, Muldowney JA 3rd, Kocalis H, Fazio S, Vaughan DE, Niswender KD. Consuming a balanced high fat diet for 16 weeks improves body composition, inflammation and vascular function parameters in obese premenopausal women. Metabolism. 2014 Apr;63(4):562-73. doi: 10.1016/j.metabol.2014.01.004. Epub 2014 Jan 17. PMID 24559846